CLINICAL TRIAL: NCT03028688
Title: HIFLO ENDO- Use of High Flow Nasal Cannula Oxygenation to Increase Patient Safety During Upper GI Endoscopy
Brief Title: HIFLO ENDO-High Flow Nasal Cannula in GI Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Anesthesia Patient Safety Foundation (Other)
Responsible Party: Principal Investigator, Michael Mazzeffi, Assistant Professor of Anesthesiology, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HP-00071111
Record Dates: First submitted 2017-01-11; First posted 2017-01-23 (Estimated); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Anesthesia Morbidity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current standard of care (No Intervention): Participants in the current standard of care will receive the usual anesthesia care for upper GI endoscopy. In addition participants will have transcutaneous PCO2 measurements performed.
- High flow nasal cannula group (Experimental): Participants in the high flow nasal cannula group will receive high flow nasal cannula oxygen and will also have transcutaneous PCO2 measurements performed.
  Interventions: Device: High flow nasal cannula oxygen

INTERVENTIONS:
Device: High flow nasal cannula oxygen — Participants will receive high flow nasal cannula oxygen delivery during anesthesia. Participants will also have transcutaneous PCO2 measurements performed using a cutaneous electrode.
  Arms: High flow nasal cannula group

SUMMARY:
Millions of patients undergo upper GI endoscopy in the United States each year. A large number of these patients have anesthesia to assist with their comfort during the procedure. The majority of patients do not have a protected airway during the procedure, meaning there is no endotracheal tube. Instead the current standard of care is to give supplementary oxygen via nasal cannula. Because patients are deeply sedated or have general anesthesia there is a risk for low oxygen saturation during the procedure, which presents a significant patient safety issue. The purpose of the clinical trial is compare the current anesthesia standard of care against high flow nasal cannula oxygen delivery during anesthesia. The investigator's hypothesis is that high flow nasal cannula oxygen delivery will decrease the frequency with which patients experience hypoxemia during anesthesia for upper GI endoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Having Upper GI endoscopy expected to last greater than 15 minutes with anesthesia.
2. Age greater than or equal to 18 years

Exclusion Criteria:

1. Propofol, midazolam, or fentanyl allergy
2. Pre-procedure plan for general anesthesia with an endotracheal tube (at the discretion of the attending anesthesiologist)
3. Any procedure with planned electro-cautery as a high-inspired oxygen concentration could increase the risk for airway or esophageal fire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Hypoxemia event (Low blood oxygen level) | The outcome variable will be measured one time 24 hours after the completion of the patient's anesthesia.
  The primary outcome measure will be occurrence of a low blood oxygen level defined by oxygen saturation less than 92% for greater than 15 seconds at any point during the patient's anesthesia. This will be a dichotomous outcome variable analyzed by time to event.

SECONDARY OUTCOMES:
Hypercarbia event (Elevated blood CO2 level) | The outcome variable will be measured one time 24 hours after the completion of the patient's anesthesia.
  The secondary outcome measure will be occurrence of an elevated blood carbon dioxide level defined as 20 mmHg above the patient's baseline value at any time during their anesthesia. This will be a dichotomous outcome variable analyzed by time to event.
Hypotension event (Low blood pressure) | The outcome variable will be measured one time 24 hours after the completion of the patient's anesthesia.
  The secondary outcome measure will occurrence of low blood pressure defined as blood pressure 25% below baseline value any time during the patient's anesthesia. This will be a dichotomous outcome variable analyzed by time to event.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Mazzeffi, MD MPH, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mazzeffi MA, Petrick KM, Magder L, Greenwald BD, Darwin P, Goldberg EM, Bigeleisen P, Chow JH, Anders M, Boyd CM, Kaplowitz JS, Sun K, Terrin M, Rock P. High-Flow Nasal Cannula Oxygen in Patients Having Anesthesia for Advanced Esophagogastroduodenoscopy: HIFLOW-ENDO, a Randomized Clinical Trial. Anesth Analg. 2021 Mar 1;132(3):743-751. doi: 10.1213/ANE.0000000000004837. PMID 32398433